CLINICAL TRIAL: NCT03960307
Title: Association of Sublingual Microcirculation Parameters and Endothelial Glycocalyx Dimensions in Resuscitated Sepsis: A Cross-sectional Study
Brief Title: Glycocalyx and Microcirculation in Sepsis
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: IDF_SDF
Record Dates: First submitted 2019-05-13; First posted 2019-05-23 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2019-05

CONDITIONS: Sepsis
Keywords: Glycocalyx; PBR; microcirculation
MeSH Terms: conditions — Sepsis | interventions — Microcirculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic patients: ICU patients with resuscitated sepsis, based on the sepsis-3 criteria. (n=30)
  Interventions: Other: Microcirculation and Glycocalyx assessment
- Healthy controls: Apparently healthy controls (n=10)
  Interventions: Other: Microcirculation and Glycocalyx assessment

INTERVENTIONS:
Other: Microcirculation and Glycocalyx assessment — Non-invasive assessment of endothelial glycocalyx dimensions (PBR) and microcirculatory parameters (e.g. PPV, PVD, TVD, MFI)

SUMMARY:
The aim of this observative, prospective study with cross-sectional design is to explore possible correlations/associations between microcirculation parameters and sublingual endothelial glycocalyx in sepsis. Therefore, 30 critically ill septic patients and 10 healthy controls were enrolled.

ELIGIBILITY:
Inclusion Criteria - septic ICU cohort:

* Sepsis (based on sepsis-3 criteria)
* ICU stay

Inclusion Criteria - healthy controls:

- Adult healthy individuals

Exclusion Criteria (for all groups):

* Underage
* pregnancy
* oral mucosal inflammation or injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Non-consecutive patients admitted in the ICU of University Hospital Münster, Germany.
  * Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Correlations between Perfused Boundary Region (PBR) and Microvascular Flow Index (MFI) measured sublingually | During ICU stay, an average of 2 days after sepsis onset
  Glycocalyx thickness will be measured with PBR (in μm) and MFI will be assessed in points. Possible correlations at a given timepoint will be explored (e.g. Spearman's Correlation).
Correlations between Perfused Boundary Region (PBR) and Proportion of Perfused Vessels (PPV) measured sublingually | During ICU stay, an average of 2 days after sepsis onset
  Glycocalyx thickness will be measured with PBR (in μm) and PPV will be assessed in percentage. Possible correlations at a given timepoint will be explored (e.g. Spearman's Correlation).
Correlations between Perfused Boundary Region (PBR) and Perfused Vessel Density (PVD) measured sublingually | During ICU stay, an average of 2 days after sepsis onset
  Glycocalyx thickness will be measured with PBR (in μm) and PVD will be assessed in mm/mm^2. Possible correlations at a given timepoint will be explored (e.g. Spearman's Correlation).

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kümpers, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- Universitiy Hospital Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rovas A, Seidel LM, Vink H, Pohlkotter T, Pavenstadt H, Ertmer C, Hessler M, Kumpers P. Association of sublingual microcirculation parameters and endothelial glycocalyx dimensions in resuscitated sepsis. Crit Care. 2019 Jul 24;23(1):260. doi: 10.1186/s13054-019-2542-2. PMID 31340868